CLINICAL TRIAL: NCT01474343
Title: An Open-label, Single Arm, Monocentric, Phase I/II Clinical Study of Intracerebral Administration of Adeno-associated Viral Vector Serotype 10 Carrying the Human SGSH and SUMF1 cDNAs for the Treatment of Sanfilippo Type A Syndrome.
Brief Title: Intracerebral Gene Therapy for Sanfilippo Type A Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LYSOGENE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1-SAF-301
Record Dates: First submitted 2011-11-10; First posted 2011-11-18 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Mucopolysaccharidosis Type III A; Sanfilippo Disease Type A
Keywords: Neurodegenerative Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Metabolic Diseases; Gene Therapy; Adenovirus Associated Vector
MeSH Terms: conditions — Mucopolysaccharidosis III; Neurodegenerative Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SAF-301 (Experimental)
  Interventions: Genetic: SAF-301

INTERVENTIONS:
Genetic: SAF-301 — The treatment plan consists on a direct injection of the investigational medicinal product SAF-301 to both sides of the brain through 6 image-guided tracks, with 2 deposits per track, in a single neurosurgical session.

SUMMARY:
The clinical trial P1-SAF-301 is an open-label, single arm, monocentric, phase I/II clinical study evaluating the tolerance and the safety of intracerebral administration of adeno-associated viral vector serotype 10 carrying the human SGSH and SUMF1 cDNAs for the treatment of Sanfilippo type A syndrome The treatment plan consists on a direct injection of the investigational medicinal product SAF-301 to both sides of the brain through 6 image-guided tracks, with 2 deposits per track, in a single neurosurgical session.

The primary objective is to assess the tolerance and the safety associated to the proposed treatment through a one-year follow up.

The secondary objective is to collect data to define exploratory tests that could become evaluation criteria for further clinical phase III efficacy studies.

Four patients will be included in the clinical trial and will be followed during one year.

The enrollment and the follow-up of the patients will take place at Bicêtre Hospital. The Neurosurgery will be performed at Necker-Enfants Malades Hospital.

Safety will be evaluating on clinical, radiological and biological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 (eighteen) months to end of 6 (six) years
* Onset of clinical manifestations related to MPSIIIA during the first 5 years of life
* SGSH activity in peripheral blood cell and / or cultured fibroblast extracts of less than 10% of controls.
* Patient affiliated to the French social security or assimilated regimens
* Family understanding the procedure and the informed consent
* Signed informed consent
* Vital laboratory parameters within normal range

Exclusion Criteria:

* Presence of brain atrophy on inclusion MRI judged on a cortico-dural distance of more than 1cm
* No independent walking (Ability to walk without help)
* Any condition that would contraindicate permanently anaesthesia
* Any other permanent medical condition not related to MPSIIIA
* Any vaccination 1 month before investigational drug administration
* Intake of aspirin within one month
* Any medication aiming at modifying the natural course of MPSIIIA given during the 6 months before vector injection
* Any condition that would contraindicate treatment with Prograf®, Modigraf®, Cellcept® and Solupred®

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Tolerance and safety | during the one year follow-up
  Measured by
  * adverse events (by type and severity)
  * clinical parameters (fever, seizure, headache, abnormal somnolence or lethargy, any new neurological symptoms),
  * radiological parameters (on MRI, any sign of bleeding after surgery, any hypersignal on T2 weighted images or diffusion images that are not at the points of injection, and any necrotic area evaluated through T1-weighted and diffusion imaging as well as modification of lipids in spectroscopy)
  * biological parameters (in particular anemia, leucopenia, thrombopenia, liver dysfunction)

SECONDARY OUTCOMES:
To collect data to define exploratory tests that could become evaluation criteria for further clinical phase III efficacy studies | during the one year follow-up
  * Brain MRI
  * Neurocognitive/behavioral tests
  * Biological markers on blood, urine and CSF

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Bicêtre - Assistance Publique des Hôpitaux de Paris, Le Kremlin-Bicêtre
  - Hôpital Necker, Assistance Publique des Hôpitaux de Paris, Paris